CLINICAL TRIAL: NCT03259568
Title: Effects of rTMS on Human Brain Activity Measured With fMRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment due to Covid-19.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00082433
Record Dates: First submitted 2017-08-15; First posted 2017-08-23 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Human Brain Activity
Keywords: TMS; BOLD activity; Network activity

STUDY DESIGN:
Intervention Model Description: The study is a within-subjects design focused on estimating the fMRI BOLD response to different levels of TMS intensity. The conditions in the study ("arms") are repeated within each participant (20%, 40%, 80%, or 120% of an individual's titrated resting motor threshold).
Who Masked: Participant
Masking Description: Participant is not informed about TMS intensity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Dose-response TMS - Intensity = 20%RMT (Experimental): Four levels of TMS intensity (here, 20% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Interventions: Device: Repetitive TMS
- Dose-response TMS - Intensity = 40%RMT (Experimental): Four levels of TMS intensity (here, 40% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Interventions: Device: Repetitive TMS
- Dose-response TMS - Intensity = 80%RMT (Experimental): Four levels of TMS intensity (here, 80% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Interventions: Device: Repetitive TMS
- Dose-response TMS - Intensity = 120%RMT (Experimental): Four levels of TMS intensity (here, 120% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Interventions: Device: Repetitive TMS

INTERVENTIONS:
Device: Repetitive TMS — 1-10 Hertz rTMS will be administered

SUMMARY:
This project investigates the effects of repetitive transcranial magnetic stimulation (rTMS) on neural circuits as a function of spatiotemporal parameters and brain state in order to better understand why the method works and how to improve its efficacy. Leveraging our expertise in application of TMS methodology during concurrent single neuron recording techniques in non-human primates and imaging and scalp potential techniques in humans, the investigators aim to resolve three interlocking problems in the design and application of rTMS: stimulation frequency, spatial targeting, and interactions with brain state.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-30.
2. Use of effective method of birth control for women of childbearing capacity.
3. Willing to provide informed consent.

Exclusion Criteria:

1. Current or recent (within the past 6 months) of substance abuse or dependence, excluding nicotine and caffeine (urine test).
2. Current serious medical illness (self report).
3. History of seizure except those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by rTMS or MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator); [TMS Adult Safety Screening (TASS) form].
4. Subjects are unable or unwilling to give informed consent.
5. Diagnosed any Axis I DSM-IV disorder (MINI, DSM-IV)
6. Subjects with a clinically defined neurological disorder including, but not limited to:

   1. Any condition likely to be associated with increased intracranial pressure
   2. Space occupying brain lesion.
   3. History of stroke.
   4. Transient ischemic attack within two years.
   5. Cerebral aneurysm.
   6. Dementia.
   7. Mini Mental Status Exam (MMSE) score of <24.
   8. Parkinson's disease.
   9. Huntington's disease.

   i. Multiple sclerosis.
7. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold.
8. Subjects with cochlear implants
9. Subjects not willing to tolerate the confinement associated with being in the MRI scanner.
10. Women who are pregnant or breast-feeding (urine test).
11. Blindness.
12. Inability to read or understand English.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active rTMS: Repetitive TMS: 1-10 Hertz rTMS will be administered, at varying levels of TMS intensity.
Period: Overall Study
Arm/Group | Active rTMS
Started | 27
Completed | 24
Not Completed | 3
Not completed — Participant performance was low | 3

BASELINE CHARACTERISTICS:
Population: Study used a within-subjects design; all 27 participants received all 4 conditions ("arms") of TMS stimulation.
Groups:
- Active rTMS (Repetitive Transcranial Magnetic Stimulation): Repetitive TMS: 1-10 Hertz rTMS will be administered, at varying levels of TMS intensity.
Arm/Group | Active rTMS (Repetitive Transcranial Magnetic Stimulation)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Within-subjects design, each subject received four TMS conditions ("arms").
  Participants
    Female | 16
    Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Within-subjects design, all conditions ("arms") were repeated in each of the 27 participants.
  Participants
    United States | 27
fMRI Activity [Mean (Standard Deviation); unit: BOLD response] — Measure reflects TMS-evoked activity associated with each TMS Intensity condition ("arm"), i.e., 20%, 40%, 80%, and 120% of an individualized resting motor threshold.
  BOLD response
    20% RMT | 1.28 (0.14)
    40% RMT | 1.28 (0.12)
    80% RMT | 1.20 (0.14)
    120% RMT | 1.25 (0.15)

OUTCOME MEASURES:

1. Primary Outcome: Motion Perception Accuracy
Description: Acute effect of a rTMS session on the performance for a motion task, as measured by accuracy (in percentage of correct responses)
Time Frame: during each TMS session, up to 3 hours
Population: Within-subjects manipulation (same subjects for each condition).
Measure: Mean (Standard Error); unit: Percentage of correct responses
Groups:
- Dose-response TMS - Intensity = 20%RMT: Four levels of TMS intensity (here, 20% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Repetitive TMS: 1-10 Hertz rTMS will be administered
- Dose-response TMS - Intensity = 40%RMT: Four levels of TMS intensity (here, 40% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Repetitive TMS: 1-10 Hertz rTMS will be administered
- Dose-response TMS - Intensity = 80%RMT: Four levels of TMS intensity (here, 80% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Repetitive TMS: 1-10 Hertz rTMS will be administered
- Dose-response TMS - Intensity = 120%RMT: Four levels of TMS intensity (here, 120% of Resting Motor Threshold), titrated to each individual, tested within the MRI.
  Outcome measures include accuracy, RT, and BOLD signal.
  Repetitive TMS: 1-10 Hertz rTMS will be administered
Arm/Group | Dose-response TMS - Intensity = 20%RMT | Dose-response TMS - Intensity = 40%RMT | Dose-response TMS - Intensity = 80%RMT | Dose-response TMS - Intensity = 120%RMT
Number analyzed (Participants) | 24 | 24 | 24 | 24
Percentage of correct responses | 63 (4.0) | 62 (4.0) | 58 (4.0) | 61 (3.0)

2. Primary Outcome: Reaction Time
Description: Acute effect of a rTMS session on the performance for a motion task, as measured by reaction time (in ms)
Time Frame: during each TMS session, up to 3 hours
Population: Within-subjects manipulation (same subjects for each condition).
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Dose-response TMS - Intensity = 20%RMT | Dose-response TMS - Intensity = 40%RMT | Dose-response TMS - Intensity = 80%RMT | Dose-response TMS - Intensity = 120%RMT
Number analyzed (Participants) | 24 | 24 | 24 | 24
milliseconds | 814 (104) | 784 (94) | 762 (85) | 810 (109)

3. Primary Outcome: Activation of Cortical Networks During a Visual Motion Task.
Description: Acute effect of a rTMS session on fMRI activation during a motion task, as measured by the change in BOLD signal
Time Frame: during each TMS session, up to 3 hours
Population: Within-subjects manipulation (same subjects for each condition).
Measure: Mean (Standard Deviation); unit: BOLD activity
Arm/Group | Dose-response TMS - Intensity = 20%RMT | Dose-response TMS - Intensity = 40%RMT | Dose-response TMS - Intensity = 80%RMT | Dose-response TMS - Intensity = 120%RMT
Number analyzed (Participants) | 24 | 24 | 24 | 24
BOLD activity | 0.89 (0.06) | 0.87 (0.05) | 0.88 (0.06) | 0.94 (0.04)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: Study used a within-subjects design; all 27 participants received all 4 conditions ("arms") of TMS stimulation.
Arm/Group | Dose-response TMS - Intensity = 20%RMT | Dose-response TMS - Intensity = 40%RMT | Dose-response TMS - Intensity = 80%RMT | Dose-response TMS - Intensity = 120%RMT
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03259568/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03259568/ICF_001.pdf